CLINICAL TRIAL: NCT04563676
Title: Physiopathology and Sequelae of COVID-19 Infection
Acronym: SEQ-COV-PHYSIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0096
Record Dates: First submitted 2020-09-23; First posted 2020-09-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Covid19; TSH; Cortisol
Keywords: Covid19; TSH; cortisol
MeSH Terms: conditions — COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood test — covid19 infected patient will have a blood test in order to make an autoimmune assessment (antinuclear antibodies, soluble nuclear anti-antigen, ANCA, antiphospholipid antibodies, FT3, FT4 , TSH, antithyroid antibodies, ACTH cortisol, and creation of a serotheque).

SUMMARY:
The data obtained from Covid-19 infections seem to suggest that the immunogenesis of Covid-19 could in some cases be the result of immune dysregulation. On the other hand, endocrine damage is possible at the tile of Covid-19 infection (mainly thyroid,adrenal, and hypothalamus). These disorders are autoimmune or linked to degeneration.

The main objective is to assess the thyroid function (thyrotropic axis) as well as the corticotropic adrenal function of patients who have had Copvid-19 pneumonia. The secondary objectives is to describe the pathophysiological mechanisms of pulmonary and vasculothrombotic involvement of Covid-19

ELIGIBILITY:
Inclusion Criteria:

* patient having a covid19 infection hospitalized at the Amiens Picardie University Hospital
* Patient who is seen in Pneumology consultation for a respiratory assessment at 3 months of his hospitalization (between M2 and M4) to evaluate presence of respiratory sequelae
* Patient who agreed to participate in the protocol
* Patient affiliated to a Social Security

Exclusion Criteria:

* patient under guardianship or curators
* patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
8-hour cortisol level in patients with Covid19 pneumonia | day 0
  8-hour cortisol level in patients with Covid19 pneumonia will be determined the day of consultation for respiratory sequelae.
TSH level in patients with Covid19 pneumonia | day 0
  TSH level in patients with Covid19 pneumonia will be determined the day of consultation for respiratory sequelae.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No